CLINICAL TRIAL: NCT02455934
Title: The Dose-response Effects of D-allulose (Psicose) With Sucrose Beverage on Glucose Tolerance and Insulin Level in Healthy Volunteers and Volunteers With Impaired Fasting Glucose
Brief Title: Effects of D-allulose (Psicose) With Sucrose Beverage on Glucose Tolerance and Insulin Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Collaborators: Kagawa University (Other)
Responsible Party: Principal Investigator, Supawan Buranapin, Assisstant Professor Supawan Buranapin, MD, Chiang Mai University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CMU-D-alloluse01
Record Dates: First submitted 2015-02-23; First posted 2015-05-28 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Impaired Glucose Tolerance
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Sucrose (Placebo Comparator): Sucrose 50 g
  Interventions: Dietary Supplement: D-allulose
- SAlloulose2.5 (Active Comparator): Sucrose 50 g + D-allulose (psicose) 2.5 g
  Interventions: Dietary Supplement: D-allulose
- SAllulose5 (Active Comparator): Sucrose 50 g + D-allulose (psicose) 5 g
  Interventions: Dietary Supplement: D-allulose
- SAllulose7.5 (Active Comparator): Sucrose 50 g + D-allulose (psicose) 7.5 g
  Interventions: Dietary Supplement: D-allulose
- SAllulose10 (Active Comparator): Sucrose 50 g + D-allulose (psicose) 10 g
  Interventions: Dietary Supplement: D-allulose

INTERVENTIONS:
Dietary Supplement: D-allulose — Eligible subjects will come for visit 1 to consume varying dose of D-allulose with sucrose beverage with 1 of 5 beverages in a random order which will be blinded for both subjects and investigators. They will have to do 24-hour dietary record a day prior to each visit. Subjects have to be abstained from energy diet within 8 hours prior to each visit. Venous blood samples will be collected 6 mL for measurement of FPG and insulin before taking any study product. Subjects have to drink all within 1 minute. Blood samples will be drawn again 6 mL at 30, 60, 90 and 120 min after consumption for measurement of PG and insulin. Every subject will be asked to come back to finish OSTT with 5 study products in a random order, each at 7 days or >5 days and <12 days apart.

SUMMARY:
Randomized, double-blind, crossover-trial, 30 subjects in each groups, either males or females, normal fasting glucose or pre-diabetes, aged > 18 years old to perform oral sucrose tolerance with either one of the 5 study products

1. Sucrose 50 g
2. Sucrose 50 g + D-allulose (psicose) 2.5 g
3. Sucrose 50 g + D-allulose (psicose) 5 g
4. Sucrose 50 g + D-allulose (psicose) 7.5 g
5. Sucrose 50 g + D-allulose (psicose) 10 g

Primary endpoints:

1. To investigate the dose-response effects of D- allulose (psicose) with sucrose beverage on glucose tolerance
2. To investigate the dose-response effects of D- allulose (psicose) with sucrose beverage on insulin levels

DETAILED DESCRIPTION:
Objectives Primary objectives

1. To investigate the dose-response effects of D-allulose (psicose) with sucrose beverage on glucose tolerance
2. To investigate the dose-response effects of D-allulose (psicose) with sucrose beverage on insulin levels

Subjects and methods Study product A. Sucrose 50 g B. Sucrose 50 g + D-allulose (psicose) 2.5 g C. Sucrose 50 g + D-allulose (psicose) 5 g D. Sucrose 50 g + D-allulose (psicose) 7.5 g E. Sucrose 50 g + D-allulose (psicose) 10 g

Study plan Screening (visit 0)

* Obtain inform consent
* History taking for medical problems, smoking, alcoholic drinking, concurrent medication, contraception or menopausal status, weight history
* Measure body weight, height and calculated BMI
* Measure waist and hip circumference
* Body composition measurement by bioelectrical impedance analysis (BIA)
* Complete physical examination
* Urine pregnancy test in all female of childbearing potential
* Provide 24-hour food record
* Ask to come back within 1 week

Visit 1: (day 7 or 6-11 days)

* Complete physical examination
* Randomize subject to receive any 1 of 5 study products
* Perform OSTT with that product
* Return food record
* Provide 24-hour food record
* Adverse events evaluation
* Ask to come back within 7 +/- 4 days

Visit 2: (day 7 or 6-11 days from visit 1)

* Complete physical examination
* Randomize subject to receive any 1 of 4 study product which are left
* Perform OSTT with that product
* Return food record
* Provide 24-hour food record
* Adverse events evaluation
* Ask to come back within 7 +/- 4 days

Visit 3 (day 7 or 6-11 days from visit 2)

* Complete physical examination
* Randomize subject to receive any 1 of 3 study product which are left
* Perform OSTT with that product
* Return food record
* Provide 24-hour food record
* Adverse events evaluation
* Ask to come back within 7 +/- 4 days

Visit 4 (day 7 or 6-11 days from visit 3)

* Complete physical examination
* Randomize subject to receive any 1 of 2 study product which are left
* Perform OSTT with that product
* Return food record
* Provide 24-hour food record
* Adverse events evaluation
* Ask to come back within 7 +/- 4 days

Visit 5 (day 7 or 6-11 days from visit 4)

* Complete physical examination
* Perform OSTT with the product that is left
* Return food record
* Adverse events evaluation

Adverse Event Assessment At each visit, participants will be asked an open question as if he/she has experienced any abnormal symptoms. Any symptom reported by the participants will be recorded as an adverse events with details of the event, its severity, start and stop dates, and relationship to study products. Gastrointestinal symptoms (heartburn, distension, nausea, vomiting, abdominal pain, flatulence, constipation and diarrhea) within 24 hours after OSTT will be asked and recorded as well.

Withdrawal criteria

1. Those who are not able to complete 5 visits of OSTT within 8 weeks
2. Those who cannot provide 24-hour dietary record at each visit
3. Those who start any medication that might cause increasing in plasma glucose during participating in the study

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age > 18 years and legal age of consent.
2. If female, the participant is either post-menopausal or surgically sterilized, or has a negative urine kit pregnancy test within 7 days prior to enrollment and will use adequate contraception during the study.
3. The participant has provided written informed consent prior to admission to the study.
4. Participant is able to join the entire study with 8 weeks.
5. Participant is able to keep 24-hour dietary record a day prior to each visit.

Exclusion Criteria:

1. Pregnancy or lactation
2. Diagnosed with diabetes mellitus
3. Those who take any medication that might be able to increase plasma glucose 1 month prior to the study or during in the study
4. Acute illness within 1 weeks prior to the study
5. Has gastrointestinal symptoms such as nausea, vomiting, loss of appetite, premature satiety, diarrhea, or chronic constipation
6. Immunocompromised status, including a debilitated state or malignancy
7. Active liver, renal, thyroid diseases
8. Lack of ability or willingness to give informed consent
9. Enrolled in any other clinical study within 3 months before enrolment
10. Any people whose life style is irregular, for example, person works at night shifts.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The dose-response effects of D-allulose (psicose) with sucrose beverage on glucose tolerance | 2 hours
  oral sucrose tolerance test with sucrose +/- allulose

SECONDARY OUTCOMES:
Time to peak plasma glucose concentration | 2 hours
  oral sucrose tolerance test with sucrose +/- allulose

OTHER OUTCOMES:
The dose-response effects of D-allulose with sucrose beverage on insulin levels after oral sucrose tolerance test | 2 hours
  Oral sucrose tolerance test with sucrose +/- allulose
Time to peak plasma insulin concentration | 2 hours
  Oral sucrose tolerance test with sucrose +/- allulose

CONTACTS AND LOCATIONS:
Overall Officials: Supawan Buranapin, MD, Principal Investigator — Chiang Mai University
Locations (1):
- Clinical trial Unit, Faculty of Medicine, Chiang Mai University, Muang, ChiangMai, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cree GM, Perlin AS. O-isopropylidene derivatives of D-allulose (D-psicose) and D-erythro-hexopyranos-2,3-diulose. Can J Biochem. 1968 Aug;46(8):765-70. doi: 10.1139/o68-117. No abstract available. PMID 4299740
- [Background] Takeshita K, Suga A, Takada G, Izumori K. Mass production of D-psicose from d-fructose by a continuous bioreactor system using immobilized D-tagatose 3-epimerase. J Biosci Bioeng. 2000;90(4):453-5. doi: 10.1016/s1389-1723(01)80018-9. PMID 16232889
- [Background] Granstrom TB, Takata G, Tokuda M, Izumori K. Izumoring: a novel and complete strategy for bioproduction of rare sugars. J Biosci Bioeng. 2004;97(2):89-94. doi: 10.1016/S1389-1723(04)70173-5. PMID 16233597
- [Background] Matsuo T, Suzuki H, Hashiguchi M, Izumori K. D-psicose is a rare sugar that provides no energy to growing rats. J Nutr Sci Vitaminol (Tokyo). 2002 Feb;48(1):77-80. doi: 10.3177/jnsv.48.77. PMID 12026195
- [Background] Matsuo T, Izumori K. d-Psicose Inhibits Intestinal alpha-Glucosidase and Suppresses the Glycemic Response after Ingestion of Carbohydrates in Rats. J Clin Biochem Nutr. 2009 Sep;45(2):202-6. doi: 10.3164/jcbn.09-36. Epub 2009 Aug 28. PMID 19794929 (Retraction: PMID 24895485 J Clin Biochem Nutr. 2014 May;54(3):219)
- [Background] Iida T, Kishimoto Y, Yoshikawa Y, Hayashi N, Okuma K, Tohi M, Yagi K, Matsuo T, Izumori K. Acute D-psicose administration decreases the glycemic responses to an oral maltodextrin tolerance test in normal adults. J Nutr Sci Vitaminol (Tokyo). 2008 Dec;54(6):511-4. doi: 10.3177/jnsv.54.511. PMID 19155592
- [Background] Hayashi N, Iida T, Yamada T, Okuma K, Takehara I, Yamamoto T, Yamada K, Tokuda M. Study on the postprandial blood glucose suppression effect of D-psicose in borderline diabetes and the safety of long-term ingestion by normal human subjects. Biosci Biotechnol Biochem. 2010;74(3):510-9. doi: 10.1271/bbb.90707. Epub 2010 Mar 7. PMID 20208358
- [Background] Hossain A, Yamaguchi F, Matsunaga T, Hirata Y, Kamitori K, Dong Y, Sui L, Tsukamoto I, Ueno M, Tokuda M. Rare sugar D-psicose protects pancreas beta-islets and thus improves insulin resistance in OLETF rats. Biochem Biophys Res Commun. 2012 Sep 7;425(4):717-23. doi: 10.1016/j.bbrc.2012.07.135. Epub 2012 Aug 1. PMID 22877751
- [Background] Ochiai M, Onishi K, Yamada T, Iida T, Matsuo T. D-psicose increases energy expenditure and decreases body fat accumulation in rats fed a high-sucrose diet. Int J Food Sci Nutr. 2014 Mar;65(2):245-50. doi: 10.3109/09637486.2013.845653. Epub 2013 Oct 21. PMID 24144428
- [Background] Matsuo T, Izumori K. Effects of dietary D-psicose on diurnal variation in plasma glucose and insulin concentrations of rats. Biosci Biotechnol Biochem. 2006 Sep;70(9):2081-5. doi: 10.1271/bbb.60036. Epub 2006 Sep 7. PMID 16960391
- [Background] Ochiai M, Nakanishi Y, Yamada T, Iida T, Matsuo T. Inhibition by dietary D-psicose of body fat accumulation in adult rats fed a high-sucrose diet. Biosci Biotechnol Biochem. 2013;77(5):1123-6. doi: 10.1271/bbb.130019. Epub 2013 May 7. PMID 23649241
- [Background] Chung YM, Hyun Lee J, Youl Kim D, Hwang SH, Hong YH, Kim SB, Jin Lee S, Hye Park C. Dietary D-psicose reduced visceral fat mass in high-fat diet-induced obese rats. J Food Sci. 2012 Feb;77(2):H53-8. doi: 10.1111/j.1750-3841.2011.02571.x. PMID 22339545
- [Background] Wong JM, de Souza R, Kendall CW, Emam A, Jenkins DJ. Colonic health: fermentation and short chain fatty acids. J Clin Gastroenterol. 2006 Mar;40(3):235-43. doi: 10.1097/00004836-200603000-00015. PMID 16633129